CLINICAL TRIAL: NCT00247741
Title: Spinal Anesthesia With Articaine and Lidocaine for Outpatient Surgery: A Double Blind Randomized Clinical Trial.
Brief Title: Spinal Anesthesia With Articaine and Lidocaine for Outpatient Surgery.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Articaine
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2005-10

CONDITIONS: Spinal Anesthesia
Keywords: spinal anesthesia; lidocaine; articaine; intrathecal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- lidocaine (Active Comparator)
  Interventions: Drug: spinal administration of lidocaine
- articaine (Experimental)
  Interventions: Drug: spinal administration of articaine

INTERVENTIONS:
Drug: spinal administration of articaine
  Arms: articaine
Drug: spinal administration of lidocaine
  Arms: lidocaine

SUMMARY:
The purpose of this study is to compare two short-acting local anesthetics, articaine and lidocaine, for spinal anesthesia in day-case surgery. The onset time of the sensory- and motor block, recovery time until discharge and complications will be studied.

DETAILED DESCRIPTION:
The ideal spinal anesthesia in day-case surgery is characterized by a short onset of sensory and motor blockade, and a rapid recovery after the operation. Short-acting local-anesthetics are used frequently in this setting.

Lidocaine is one of the agents that is used most frequently. It has been associated with an increased incidence of Transient Neurological Symptoms (TNS). Articaine is another agent that is being used more often and is said to act faster and shorter than lidocaine.

We will compare spinal anesthesia with lidocaine and articaine in a randomized double-blind clinical trial. Endpoint are:

* onset of sensory and motor block
* recovery from sensory and motor block
* time to micturition
* patient satisfaction
* complications

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* ASA I-III
* Patients planned for a short surgical procedure on lower extremities or lower abdomen.
* Procedure in day-case setting
* Procedure under spinal anesthesia
* Informed consent

Exclusion Criteria:

* Contra-indications spinal anesthesia
* History of allergic reactions on amide-type local anesthetics
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2005-11; Study Completion 2006-05

PRIMARY OUTCOMES:
Onset time (sec) of sensory and motor blockade (after administration of drug)
Recovery time (min) from sensory and motor blockade
Spread of sensory blockade (30 min after administration of drug, dermatomal level)

SECONDARY OUTCOMES:
Hemodynamic stability (lowest systolic blood pressure, vasopressor therapy)
Complications
Patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Leon Timmerman, MD, Principal Investigator — St Antonius Hospital, dept. of anesthesiology; Emile MJ Andriessen, MD, Study Chair — St Antonius Hospital, dept of anesthesiology
Locations (1):
- St Antonius Hospital, Nieuwegein, Utrecht, Netherlands

REFERENCES:
- [Background] Vree TB, Gielen MJ. Clinical pharmacology and the use of articaine for local and regional anaesthesia. Best Pract Res Clin Anaesthesiol. 2005 Jun;19(2):293-308. doi: 10.1016/j.bpa.2004.12.006. PMID 15966499
- [Result] Kaukinen S, Eerola R, Eerola M, Kaukinen L. A comparison of carticaine and lidocaine in spinal anaesthesia. Ann Clin Res. 1978 Aug;10(4):191-4. PMID 360957